CLINICAL TRIAL: NCT03519191
Title: Healthy Relationships and Economic Pathways Evaluation Study
Brief Title: Healthy Relationships and Economic Pathways
Acronym: H-REP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment too low for power analysis
Sponsor: Public Health Institute, California (Other)
Collaborators: American Institutes for Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PHICalifornia
Record Dates: First submitted 2018-04-06; First posted 2018-05-08 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Adolescent Relationship Abuse; Sexually Transmitted Infections; Pregnancy (Unwanted); Violence; Intentional Injury
Keywords: teen dating violence; sexual assault; reproductive coercion
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: This socio-behavioral intervention project will randomly assign participants to the HRE-only or the HRE+Technology bootcamp arms, with a waitlist for accommodation of additionally interested youth, and a cross-over option
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Relationships Education (HRE) (Other): Social-behavioral intervention Participants will receive employment support services and Healthy Relationships Education interventions.
  Interventions: Behavioral: Healthy Relationships Education (HRE)
- HRE+Technology Bootcamp (Other): Social-behavioral intervention + technology bootcamp (associated economic pathways for participants) Participants will receive employment support services, Healthy Relationships Education, and Technology Bootcamp interventions.
  Interventions: Behavioral: HRE+Technology Bootcamp

INTERVENTIONS:
Behavioral: Healthy Relationships Education (HRE) — Healthy Relationships and Economic Pathways involves formal classes in Healthy Relationship Education (HRE), comprehensive case management, and support services and referrals to services.
  Arms: Healthy Relationships Education (HRE)
Behavioral: HRE+Technology Bootcamp — HRE + Technology Bootcamp involves formal classes in Healthy Relationships Education (HRE), comprehensive case management, support services and referral to services, 6-week intensive website and professional development training, and paid work experience developing a website for a local small business and mentorship.
  Arms: HRE+Technology Bootcamp

SUMMARY:
The California Adolescent Health Collaborative (CAHC) brings together multiple nonprofit organizations in California's Central Valley to implement the Healthy Relationships and Economic Pathways (H-REP) program, which aims to increase and promote healthy relationships and stability among youth between the ages of 14 and 24.

DETAILED DESCRIPTION:
This research project was designed to explore three core questions (RQs).

Research Question 1:Does assignment to the HRE improve the knowledge and skills necessary to develop and maintain caring and supportive personal and professional relationships among youth between the ages of 18 and 24 in Stanislaus and Merced Counties?

In addition, American Institutes for Research (AIR), an independent evaluator, has been asked to answer two supplemental RQs:

Research Question 2: Does participation in the HRE Technology Boot Camp improve technological knowledge and skills as well as awareness of professional and educational opportunities among youth between the ages of 18 and 24?

Research Question 3: Does HRE have the same effect on relationship knowledge and skills for youth between the ages of 18 and 24 who participate in the HRE-only training as it does for youth who participate in HRE plus Technology Bootcamp?

H-REP provides a comprehensive, three-pathway program of services to (a) students in traditional, comprehensive high schools; (b) students in continuation of alternative schools (e.g. court schools); and (c) youth between the ages of 18 and 24 who are receiving employment support services from Central Valley nonprofit programs. The H-REP program involves formal classes in Healthy Relationship Education (HRE) and technology use, case management, and job skills training.

ELIGIBILITY:
Inclusion Criteria:

* students in traditional, comprehensive high schools; students in continuation or alternative schools; youth between ages of 18-24 who receive employment support services from Central Valley non-profit programs (California); residents of Merced or Stanislaus counties (California).

Exclusion Criteria:

* less than sixth-grade English language proficiency

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
HRE survey to assess changes in knowledge and skills needed to develop and maintain caring and supportive personal and professional relationships (surveys) | 6 months
  Baseline and 6 month follow-up surveys of participants will be conducted to assess impact of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Chopel, DrPH, Principal Investigator — Public Health Institute
Locations (1):
- Public Health Institute, Oakland, California, United States